CLINICAL TRIAL: NCT04414319
Title: Impact of SARS-CoV-2 Infection in a Population Aged 70 Years or Older on Loss of Autonomy
Brief Title: Severe Acute Respiratory Syndrome-Coronavirus-2 and Loss of Autonomy in the Elderly
Acronym: CovAged
Status: Terminated | Type: Observational
Why Stopped: Lack of time to realize the research
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 20_RIPH3-02
Record Dates: First submitted 2020-05-18; First posted 2020-06-04 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: SARS-CoV 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In most diseases, older people have less typical symptomatology than that described for younger people. The investigators therefore hypothesize that within the framework of coronavirus disease 19, the clinical pictures in the elderly will present specificities that will need to be described. Moreover, since infection by the severe acute respiratory syndrome (SARS-CoV-2) virus is new to humans, the investigators do not yet have sufficient information on the fate of the elderly, in terms of loss of autonomy, rehospitalization, institutionalization, mortality, etc. the investigators therefore assume that the clinical pictures in the elderly will present specificities that will need to be described. The investigators hypothesize that an acute infection of this type will have short-, medium-, and long-term repercussions in the elderly.

DETAILED DESCRIPTION:
The question of the outcome of elderly populations in the immediate aftermath of the epidemic and at a distance from it are essential to measure the effectiveness of the medical care that has been undertaken, but also to adapt the response to the specific problems of the elderly population. It is likely that the older, more fragile population will take longer to recover from the epidemic than the younger population because their functional reserves prior to coronavirus disease 19 are lower. In addition, the possible consequences of containment must be added to the burden of co-morbidities and dependence prior to the epidemic. Containment is synonymous with a restriction in social relationship, and sometimes a reduction in the support provided on a daily basis to frail or even dependent elderly people. Moreover, containment alone may be responsible for the onset or worsening of pathologies.

In most diseases, older people have less typical symptomatology than that described for younger people. The investigators therefore hypothesize that within the framework of coronavirus disease 19, the clinical pictures in the elderly will present specificities that will need to be described. Moreover, since infection by the SARS-CoV-2 virus is new to humans, the investigators do not yet have sufficient information on the fate of the elderly, in terms of loss of autonomy, rehospitalization, institutionalization, mortality, etc. The investigators therefore assume that the clinical pictures in the elderly will present specificities that will need to be described. The investigators hypothesize that an acute infection of this type will have short-, medium-, and long-term repercussions in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older;
* Hospitalized in a short stay or a rehabilitation geriatric wards at one of the participating centers;
* Positive by Reverse Transcriptase-Polymerase Chain Reaction for severe acute respiratory syndrome (SARS-CoV-2) coronavirus or be considered to have SARS-CoV-2 coronavirus based on lung CT data and physician opinion;
* Formal consent to answer the questionnaire or, in the event of inability to give consent, consent obtained from the trusted third party;
* Affiliation to a social security scheme.

Exclusion Criteria:

* Patient under formal guardianship or trusteeship.

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: A cohort of covid-19 patients aged 70 years or older, admitted in a short stay or a rehabilitation geriatric wards.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Loss of autonomy | 36 months
  Loss of autonomy (based on the variation of activity of daily living and instrumental activities of daily living score, and new formal or informal help)

SECONDARY OUTCOMES:
Hospital readmission | 1 month follow-up
  Any new hospitalization not scheduled during follow-up. We we will also study early re-hospitalizations (occurring within 30 days or less).
Nursing home admission | 36 months
  for non-institutionalized persons at inclusion) by a change of residence, from the usual place of residence to a lodging establishment for people dependent elderly, or to a long-term care unit
All-cause mortality | Inclusion and 36 months
  Death considered will be those occurring between inclusion and the end of follow-up
change in self-rated health | 36 months
  Self-rated health will be rated as: very good, good bad, very bad. The transition during monitoring to a less favorable modality than that announced at inclusion will be considered as a perceived deterioration in health

CONTACTS AND LOCATIONS:
Overall Officials: Moustapha DRAME, PHD, Study Director — Unversity hospital of Martinique
Locations (5):
- France (3):
  - University hospital of Rennes, Rennes
  - Va de Lys-Ramsay Gds group Clinic, Tourcoing
  - Hopsital of Valenciennes, Valenciennes
- University hospital of Guadeloupe, Les Abymes, Guadeloupe
- University hospital of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No